CLINICAL TRIAL: NCT00400348
Title: A Phase 2, Open-Label, Safety and Efficacy Study of Panzem® Nanocrystal Colloidal Dispersion Administered Orally in Patients With Recurrent or Resistant Epithelial Ovarian Cancer
Brief Title: Safety and Efficacy Study of Panzem® Nanocrystal Colloidal Dispersion in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Chief Medical Officer, EntreMed, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-CLN-004
Record Dates: First submitted 2006-11-14; First posted 2006-11-16 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

INTERVENTIONS:
Drug: Panzem Nanocrystal Colloidal Dispersion (NCD) — Panzem NCD 1,000 mg, four times daily for 28 consecutive days

SUMMARY:
The purpose of this study is to evaluate the efficacy, limited pharmacokinetics (PK), and safety of 1,000 mg of Panzem® NCD administered orally four times a day to patients with recurrent or resistant epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of protected health information.
2. Have histologically-confirmed:

   * epithelial ovarian cancer or
   * primary peritoneal carcinomatosis or
   * fallopian tube cancer. Enrollment of patients with clear cell histology is encouraged.
3. Have measurable disease according to RECIST or detectable disease by 1) CA-125 at least twice the ULN within 14 days prior to registration for protocol therapy; 2) Ascites and/or pleural effusion attributed to tumor; 3) solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST definitions for target lesions. Radiographic assessments must be obtained within 28 days prior to registration for protocol therapy.
4. Be 18 years of age or older at the time of consent.
5. Be at least 4 weeks since last anti-cancer treatment, radiation or surgery at the time of registration for protocol therapy (with the exception of hormonal therapy, where a 1 week wash-out period is sufficient; minor surgeries, such as catheter placement or removal within 1 week from enrollment are allowed).
6. Have failed at least one prior platinum based chemotherapeutic regimen. (Platinum failure is defined as Platinum-refractory (progression while receiving a platinum-containing regimen) or platinum-resistant (disease progression within 6 months from completion of platinum-containing regimen).
7. Have life expectancy of at least 3 months.
8. Have ECOG performance status of 0 or 1 as assessed within 14 days prior to registration for protocol therapy.
9. Have near-normal organ function, as evidenced by laboratory data within 14 days prior to registration for protocol therapy:

   * Aspartate aminotransferase and alanine aminotransferase less than 2.5 times upper limit of normal (ULN)
   * Total bilirubin less than 1.5 times ULN
   * Alkaline phosphatase less than 2.5 times ULN
   * Absolute neutrophil count greater than or equal to 1,500 cells/mm3
   * White blood cell count greater than or equal to 3,000 cells/mm3
   * Hemoglobin greater than or equal to 9.0 g/dL
   * Platelets greater than 75,000/mm3
   * Creatinine levels less than 1.5 times ULN
10. Have no evidence of bowel obstruction, malabsorption, or other contraindication to oral medication.
11. Females of childbearing potential must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) while on treatment.
12. Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy. Subjects are considered not of childbearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.

Exclusion Criteria:

1. Be breastfeeding.
2. Have any condition that is likely to interfere with regular follow-up.
3. Have a history of myocardial infarction or angina pectoris or angina equivalent within 6 months prior to registration for protocol therapy (the patient may be on anti-anginal medications if the symptoms can be entirely controlled), or have uncontrolled hypertension or congestive heart failure.
4. Have participated in any clinical trial involving conventional or investigational drugs or devices within 4 weeks prior to registration for protocol therapy.
5. Have had any active cancer in addition to the epithelial ovarian cancer within the last 5 years, with the exception of:

   * superficial skin cancer (basal cell or squamous cell skin carcinoma)
   * carcinoma in situ of the cervix
   * Stage I endometrial cancer with less than 50% invasion of the myometrium, or
   * other adequately treated Stage I or II cancer in complete remission.
6. Have an active infection requiring antibiotic treatment.
7. Be receiving concurrent anticoagulation therapy (low dose coumadin for port-a-cath maintenance is allowed).
8. Have any additional uncontrolled serious medical condition or psychiatric illness.
9. Be receiving combination anti-retroviral therapy for the treatment of immunodeficiency.
10. Have brain metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Assess the safety of oral doses of Panzem NCD administered to patients with recurrent epithelial ovarian cancer | Throughout study participation

CONTACTS AND LOCATIONS:
Overall Officials: Daniela E. Matei, M.D., Study Chair — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States